CLINICAL TRIAL: NCT04267835
Title: Prospective Cohort Study on Mid-term Safety and Effectiveness of Minimal Invasive Coronary Artery Bypass Grafting
Brief Title: Prospective Cohort Study on Minimal Invasive Coronary Surgery
Acronym: PCSMICS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKU MICS study
Record Dates: First submitted 2019-05-19; First posted 2020-02-13 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Bypass, Off-Pump
Keywords: Coronary artery bypass grafting; Minimally Invasive Surgical Procedures; Off-pump CABG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MICS (Minimal invasive coronary surgery): Patients undergoing MIDCAB surgery.
  Interventions: Procedure: MIDCAB
- OPCABG (thoracotomy off-pump CABG): Patients undergoing thoracotomy OPCABG surgery
  Interventions: Procedure: thoracotomy OPCABG

INTERVENTIONS:
Procedure: MIDCAB — Surgery: MIDCAB
  Groups: MICS (Minimal invasive coronary surgery)
Procedure: thoracotomy OPCABG — Surgery: thoracotomy OPCABG
  Groups: OPCABG (thoracotomy off-pump CABG)

SUMMARY:
CABG technology is recognized as the preferred treatment, and its major adverse cardiac and cerebral event(MACCE) incidence and mortality are lower than percutaneous coronary intervention(PCI). However, the traditional CABG procedure requires sternal incision, large trauma and long recovery period after surgery.

How to reduce trauma and treat multiple complex coronary lesions under minimally invasive conditions has become a hot spot. MIDCAB surgery can complete the coronary anastomosis only by a 6-8 cm incision in the left chest. It has been more than ten years since the first literature report in the world, however, due to the technical bottleneck, a unified and standardized surgical procedure has not yet been formed. Some centers are still in the exploratory stage, and internationally Large-scale studies of clinical outcomes (mostly less than 150 cases) have not been reported. Assessing the minimally invasive procedure's safety and effectiveness has become an urgent problem to be solved.

At present, our center has completed nearly 200 cases of small incision multi-coronary coronary artery bypass graft surgery. The investigators evaluate the patency of the graft by the postoperative of angiography, the patency of grafts is more than 95%, and there is no statistical difference with conventional OPCABG. On the other hand, focus on the postoperative complications, there was no significant difference in the incidence of MACCE and revascularization between the MIDCAB group and conventional surgery during hospitalization. The investigators assume that the early results of this procedure are safe and effective. MIDCAB has a congenital advantage because of its' reduction of the trauma of the thoracotomy and the aesthetics of the incision. Therefore, if a larger sample size study and mid-term follow-up results are obtained, and the conclusion prove that the safety of the small incision surgery and the patency of the grafts are not inferior to conventional surgery. The investigators can consider that minimal invasive coronary surgery(MICS) is a technique worth trying to promote.

Through this prospective cohort study, the investigators evaluated the safety of MICS through mid-term follow-up results and asses the efficiency by the results of grafts patency (angiography or CT within 30 days after surgery) and medical outcomes study-short from scores(SF-36), establish the surgical standard and perioperative management method.

DETAILED DESCRIPTION:
1. MIDCAB procedure introduction

   1. Surgery preparation:

      General anesthesia, double lumen tracheal intubation. In the supine position, tilt 15° to the right. An automatic defibrillation electrode is attached to the right front and left rear chest wall, and the external defibrillator is connected. A small incision of 8-10 cm into the left anterior lateral 5th intercostal space was performed into the chest.
   2. Internal mammary artery acquisition:

      After entering the chest, the IMA is exposed through a new minimal invasive retraction system. Single or bilateral IMA is obtained as needed. Separate the IMA From the middle segment (non-fat muscle coverage area) applied with an electric scalpel (15J), and the free range was up to the first rib to the fifth or sixth intercostal(IMA bifurcation).
   3. Bypass strategy:

      All procedures were performed under a non-cardiopulmonary situation, and vascular anastomosis was performed with the aid of a laparoscopic cardiac stabilizer. The stabilizer is smaller and does not occupy the operating space. The head of stabilizer can be rotated 360 degrees and the target vessel can be fixed at any angle. Bilateral internal mammary artery, radial artery and saphenous vein can be used as graft vessels. The bypass strategy is not particularly different from conventional bypass surgery, including aorta(AO)-saphenous vein graft (SVG) or radial artery(RA)-X1-X2-...( sequential anastomosis), left internal mammary artery(LIMA)-right internal mammary artery(RIMA) -RA or SVG(Y)-X, RIMA-left anterior descending(LAD), LIMA-RA or RIMA or SVG(I)-X1-X2 and so on.
   4. Vascular anastomosis:

      The target vessel is exposed through the pericardial suture, the heart is locally fixed with the aid of a cardiac stabilizer, and the target vessel is inserted shunt to avoid hemodynamic disorder and arrhythmia. Vascular anastomosis is performed by 8-0 polypropylene suture.
   5. Aortic exposure and proximal anastomosis:

      Place gauze behind the aorta, expose the aorta with the right pericardial suspension suture, temporary block aortic anterior wall with a soft-chain sidewall clamp, Punch on the aortic anterior wall with 3.5mm puncher, anastomose SVG or RA on AO with 6-0 polypropylene suture.
   6. postoperative management: Patients go to the cardiac ICU ward postoperatively. The investigators closely observe the electrocardiogram and myocardial enzyme changes, maintain a mean arterial pressure more than 70 mmHg perfusion pressure, and the use of nitrate ester drug to relax coronary, Begin with oral aspirin (100 mg, qd) antiplatelet therapy as soon as tracheal intubation is removed. Complete chest X-ray, cardiac ultrasound and coronary angiography before discharge.
   7. Patient selection Because MIDCAB requires the heart to be exposed through the lateral incision, it is necessary to avoid the difficulty of exposure caused by thoracic deformity, adhesion or obesity; it is not suitable for MIDCAB in patients with extremely low cardiac function and severe heart enlargement; Because of the necessity of single-side ventilation, such as patients with severe pulmonary dysfunction before surgery, should also avoid small incision surgery. See the eligible and exclusion criteria for details.
2. Baseline matching problem MIDCAB is more rigorous in terms of patient selection, such as weight, EF%, and lung function, thus the study will use a propensity score method to match the baseline of two groups to eliminate the baseline bias.

   Baseline factor： General: gender, age, BMI History and comorbidities：Smoke, Diabetes (diagnostic criteria: oral hypoglycemic agents, insulin therapy, HbA1c greater than 7.0%, postprandial blood glucose greater than 11.1mmol/L, fasting plasma glucose greater than 7.0mmol/L), previous stroke(CT showed large area softening lesion) and presence of neurological dysfunction (paralysis, weak muscles, aphasia, paresthesia, and difficulty urinating), Hyperlipidemia (administered or admitted to hospital serum cholesterol greater than 5.17mmol / L or 200mg / dl), high blood pressure (blood pressure greater than 140 / 90 mmHg without medication), renal insufficiency (dialysis or serum creatinine level greater than 140mmol / L ), Peripheral vascular disease (preoperative ultrasound or CT confirmed peripheral vascular stenosis greater than 50%), previous history of cardiac surgery, previous PCI history (balloon dilatation or stent implantation)

   Preoperative status: Classification of angina (stable angina pectoris, unstable angina pectoris, non st-t segment elevation myocardial infarction, st-t segment elevation myocardial infarction), previous myocardial infarction history(pathological Q wave on ECG, abnormal segment motion on lesion area accompany with low EF% or clear and definitely evidence of elevation of creatine kinase(CK-MB) or troponin(cTnI), New York Heart Association(NYHA) heart function classification.

   Preoperative examination:creatinine(Cr), N-terminal pro brain natriuretic peptide(NT-proBNP), total cholesterol(TG) and low density lipoprotein(LDL) level, preoperative cardiac function (EF%, LVEDmm), SYNTAX score (evaluation by cardiologist).

   Preoperative medication (within 1 week): aspirin, clopidogrel
3. statistical methods The primary endpoint of 12 months MACCE will be analysis by non-inferiority method. The small incision surgery has advantage of little trauma and the aesthetics of the incision. According to the results of previous studies and literature reports, the 1 year graft's patency is assumed to be 96% in the MICS group, 96% in the control group, test performance β=90%, in the single-tail test α=0.025, △=0.06, the investigators expected the sample size of each group is required to be 168, and assume drop rate is about 15%, and finally 190-200 cases are needed in each group. In the OPCABG group, considering the propensity score matching efficiency of 0.5, it may be need more cases.

The other primary endpoints of Physical Component Scale (PCS) will be analysis by superior effect test. The higher the PCS score of SF-36 scale, the better the patient's physiological health. According to previous studies and literature reports, the average PCS score of SF-36 scale on the 30th day after CABG was 43 with a standard deviation of 10. The PCS difference of SF-36 scale with the smallest clinical significance reported in literature was 2. Through previous studies, the average PCS score on the 30th day after CABG in MICS group was 50. Assuming that the lower line of 95% confidence interval of PCS score difference between MICS-CABG group and OPCABG group is greater than 2, it is considered that the PCS score of MICS-CABG group is better than OPCABG group, with inspection level α=0.025 (one side) and inspection efficiency 1-β=0.80. The sample size of OPCABG group and MICS group is calculated to be 65 cases, with an estimated miss rate of 20%, and each group needs to include at least 82 people.

Based on the above conclusions, The investigators calculated sample size is 200 cases in each group.

After establishing the database, the logistic regression model will be established，the dependent variable is surgery procedure（MICS surgery）, the independent variable are baseline factor, and the receiver operating characteristic curve(ROC) will be drawn. The logistic regression model will be used to calculate the prone score(PS) of each subject. The nearest neighbor matching method will be used to select the thoracotomy OPCABG cases in a 1:1 ratio according to the priority matching method.

According to the basic principles of Intention-to-Treat (ITT), the whole analysis set was used. The analysis of the main indicators will include all randomized subjects, whether or not they will complete the test, the data will be included in the analysis.

Statistics data include baseline analysis, primary endpoints, secondary endpoints, observations, and compliance indicators. Measurement data that conformed to the normal distribution will be statistically described using mean ± standard deviation (χ ± S，using t test). Non-normally distributed measurement data will be statistically described using median and quartiles (using variance or nonparametric tests). The grade data will be tested using rank sum test. The count data will be statistically described as a percentage, and two or more independent sample rates will be compared using a chi-square test. Fisher's exact probability analysis will be used for indicators with low index positives (expected value <5). Survival-related data will be applied by proportional hazards model(COX) regression and survival curve risk.

Describe the missing value processing method: The estimation of the missing value of the main indicator is carried forward using the closest observation when selecting the full analysis set for statistical analysis,

5、 Ethics and safety Ethics: This research has been reviewed and filed by the Ethics Committee of the Third Hospital of Peking University. Informed consent will be signed before each participating patient was enrolled Safety: Through pre-research, MICS is a safe and effective new surgical procedure. At present, the investigators have completed more than 200 MICS operations. Only 2 of these patients died, and the postoperative complications and mid-term follow-up results were counted. The rate of graft patency and complications is not inferior to thoracotomy OPCABG surgery.

6、 Quality control Access system: MICS surgery is limited by the operation space. Although the multiple minimal invasive bypass surgery can be achieved routinely at present in our center, this surgery requires high skill and long learning curve. The cardiac surgery will strictly implement the surgeon's access qualification and have regular bypass surgery 300. For example, in the case of a small incision, only 50 patients with more than one bypass surgery, after a discussion within the department and approved by the core group, can perform small incision multi-bridge surgery.

Safeguard plan: For each case of small incision surgery, the patient's clinical data will be evaluate preoperative in our center by more than 3 senior surgeons. The surgical plan is strictly according to the standard of admission; Femoral arteriovenous will be routinely prepared for emergency cardiopulmonary bypass(CPB) and intraaortic balloon pumping(IABP) implantation. Transformation to thoracotomy surgery will be carried out if hemorrhage, uncontrollable hemodynamic disorder and malignant arrhythmia occured.

Termination of research criteria:

To ensure the safety of all candidates, a quality and safety management team will be established to monitor the complications and major safety indicators of the MICS group. The data were collected monthly to monitor serious complications (death, MACCE, unplanned revascularization, reoperation etc.) Our research will be terminated when any of the serious complications happen more than 5 cases .

ELIGIBILITY:
Inclusion Criteria:

Patients are planned for undergoing off-pump coronary artery bypass surgery.

Exclusion Criteria:

1. BMI greater than 28
2. trauma, surgical or radiotherapy history of left chest
3. EF less than 40%
4. Simultaneous other cardiac surgery or planned cardiopulmonary bypass
5. Preoperative critical situation: acute myocardial infarction, heart failure and other conditions require emergency surgery. Preoperative nitrate drugs are difficult to control angina and needs IABP implantation.
6. Respiratory function: severe hypoxemia (pO2 less than 60 mmHg without Oxygen inhalation), carbon dioxide retention (pCO2 > 50 mmHg), severe chronic obstructive pulmonary disease (FEV1/forced vital capacity less than 70% and FEV1 less than 50%)
7. Aortic lesions: patients with ascending aorta calcification confirmed by preoperative CT
8. Peripheral vascular lesions:By the preoperative assessment with ultrasound or CT，LIMA and left subclavian artery stenosis>70% ,or bilateral femoral artery calcification, stenosis>50%
9. Drug therapy: Preoperative antiplatelet or anticoagulant therapy (except aspirin and clopidogrel)
10. Others: Exclusion criteria and contraindications of CABG

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are planned for undergoing off-pump coronary artery bypass surgery.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of 1 years graft occlusion rate | 12 months after the MIDCAB or OPCABG surgery
  12 months occlusion rate of graft(Evaluate by angiography of CT angiography )
30 days PCS scores | 30days after the MIDCAB or OPCABG surgery
  PCS scores calculated from the SF-36
30 days mental health summary scales(MCS) of SF-36 scores | 30days after the MIDCAB or OPCABG surgery
  MCS scores calculated from the SF-36

SECONDARY OUTCOMES:
Rate of 30 days graft occlusion rate | within 30days after the MIDCAB or OPCABG surgery
  perioperative occlusion rate of graft(Evaluate by angiography of CT angiography )
MCS scores | 7 days, 3 months, 6 months and 12 months after the MIDCAB or OPCABG surgery
  MCS scores calculated from the SF-36
PCS scores | 7 days, 3 months, 6 months and 12 months after the MIDCAB or OPCABG surgery
  PCS scores calculated from the SF-36
Rate of Perioperative MACCE | Within 30 days of the MIDCAB or OPCABG surgery
  Major adverse cardiovascular and cerebrovascular events（ Composite endpoint of Myocardial infarction, Stroke and death)
Rate of mid-term MACCE incidence | 12 months after the MIDCAB or OPCABG surgery
  Major adverse cardiovascular and cerebrovascular events（ Composite endpoint of Myocardial infarction, Stroke and death)

OTHER OUTCOMES:
Number of Transfusion volume | Within 30 days after the MIDCAB or OPCABG surgery
  Perioperative transfusion number(U) of red blood cell
mechanical ventilation time (hours) | Within 30 days after the MIDCAB or OPCABG surgery
  Perioperative mechanical ventilation time
Rate of wound infection | Within 90 days of the MIDCAB or OPCABG surgery
  wound infection performed as redness, exudation, cracking, delayed healing that need surgical suture
Rate of secondary surgery | Within 30 days after the MIDCAB or OPCABG surgery
  All cause secondary surgery event such as bleeding, hemodynamic instability, sternum fracture or wound infection etc.
Rate of other complications | Within 30 days after the MIDCAB or OPCABG surgery
  Renal failure、atrial fibrillation、postoperativeIABP implantation、postoperative extracorporeal membrane oxygenation(ECMO) implantation etc.
Rate of Perioperative mortality | Within 30 days of the MIDCAB or OPCABG surgery
  all cause death no matter cardiogenic death or non-cardiogenic death
Rate of Mid-term mortality | Within 12 months after the MIDCAB or OPCABG surgery
  all cause death no matter cardiogenic death or non-cardiogenic death
Rate of Revascularization | Within 12 months after the MIDCAB or OPCABG surgery
  Receive PCI or Redo-CABG because of graft stenosis or occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Ling, Doctor, Study Chair — Peking University Third Hospital; Yichen Gong, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding T, Gong Y, Fu Y, Cui Z, Wu S, Yang W, Yang H, Zhao H, Feng H, Zheng H, Meng L, Guo R, Han H, Ling Y. Minimally invasive coronary bypass grafting for treating multivessel coronary disease: A single-center prospective pilot study. JTCVS Open. 2025 May 4;25:96-119. doi: 10.1016/j.xjon.2025.03.030. eCollection 2025 Jun. PMID 40631015